CLINICAL TRIAL: NCT00878371
Title: Identification and Quantification of the Effects of a Surgery-induced Peripheral Inflammatory Response on Changes in Drug Efflux Transporter Function in the Brain
Brief Title: Effects of a Surgery-induced Peripheral Inflammatory Response on the Blood Brain Barrier
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Richard Hall, MD FRCPC FCCP, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hall Morphine TAA-01
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Dissecting Aneurysm of the Thoracic Aorta
Keywords: morphine; blood brain barrier; surgery induced peripheral inflammatory response
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- morphine (Other): All patients treated with Morphine during induction after the lumbar drain inserted. Morphine was prescribed as Standard of care post operatively
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: morphine — All patients treated with Morphine during induction after the lumbar drain inserted. Morphine was prescribed as Standard of care post operatively

SUMMARY:
The purpose for this study is to determine if surgery (repair of descending thoracic aneurysm) causes a temporary decrease in the Blood Brain Barrier's ability to remove drugs from the brain back into the blood. The Blood Brain Barrier surrounds the brain and the spinal cord. This Blood Brain Barrier acts as a filter and allows some things to cross into the brain and allows other matter to be removed. Studies have shown the Blood Brain Barrier is affected by inflammation.

Functions of the Blood Brain Barrier in animals have been studied. Human studies with multiple causes of inflammation (e.g. Alzheimer's, Epilepsy, trauma and severe infections in critically

Hypothesis: Surgically-induced inflammation will temporarily reduce blood-brain barrier drug efflux transporter function in proportion to the degree of inflammation. The investigators anticipate that inflammation-mediated reductions in drug transporter function will be reflected by an increased cerebral spinal fluid (CSF) concentration of morphine (a PGP substrate) and M3G and M6G (MRP1 substrates). The corresponding in vitro studies will allow us to elucidate the mechanism(s) by which inflammation alters blood brain barrier efflux transport of morphine, M3G and M6G.

DETAILED DESCRIPTION:
Study Objectives: To determine the role of surgery-induced inflammation on the transport of morphine and its metabolites, M3G and M6G, across the blood-brain barrier.

Study phase: IV Study Design: This is a sequential enrolment study design in which elective surgical patients presenting for repair of an ascending thoracic aneurysm and fitted with a CSF drain as part of their standard of care will be approached for permission to draw blood samples at specified times during their hospital course. Concomitantly, samples of CSF will be collected from the CSF drainage system (CSF is normally wasted).

Morphine will be used as the primary analgesic agent (this is within the standard of care). Samples will be collected at specified time intervals for 5 days or until the CSF drain is removed (whichever comes first). Samples collected will be analysed for morphine, its 3- and 6- glucuronide metabolites, inflammatory cytokines, markers of CNS injury and anatomical integrity of the BBB. Area under the concentration vs. time curve will be calculated and the effect on morphine metabolism and penetration across the BBB will be determined using a repeated measures analysis of variance technique (as used in our previous study).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are to undergo elective surgery for thoracic aortic vascular disease requiring insertion of a lumbar CSF drain
2. Informed consent will be obtained from the subject or authorized legal representative -

Exclusion Criteria:

1. Unwilling or unable to provide informed consent
2. Sensitivity or documented allergy to morphine
3. Inability to place lumbar CSF drain
4. Dialysis dependent -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome variables are the correlation between the ratio of CSF/plasma morphine , morphine-3-glucuronide (M3G), and morphine-6-glucuronide (M6G) levels and the plasma concentration of IL-6 over time. | CSF and Blood samples will be taken in the OR, post operatively ( every 6 hrs until POD 5 if CSF drain still in place)

SECONDARY OUTCOMES:
Correlation between CSF/Plasma ratios of morphine, M3G, M6G and plasma concentration of TNFα and ET-1 over time. | CSF and Blood samples will be taken in the OR, post operatively ( every 6 hrs until POD 5 if CSF drain still in place)
Correlation between CSF/plasma ratios for morphine, M3G, M6G and CSF/Plasma ratios for albumin and S-100β over time. | CSF and Blood samples will be taken in the OR, post operatively ( every 6 hrs until POD 5 if CSF drain still in place)

CONTACTS AND LOCATIONS:
Overall Officials: Richard I Hall, MD, Principal Investigator — Capital Health- Queen Elizabeth II Health Sciences Center
Locations (1):
- Capital Health- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
publication in process

REFERENCES:
- [Background] Roberts DJ, Goralski KB. A critical overview of the influence of inflammation and infection on P-glycoprotein expression and activity in the brain. Expert Opin Drug Metab Toxicol. 2008 Oct;4(10):1245-64. doi: 10.1517/17425255.4.10.1245. PMID 18798696
- [Derived] Roberts DJ, Hall RI, Wang Y, Julien LC, Wood J, Goralski KB. S100B as a biomarker of blood-brain barrier disruption after thoracoabdominal aortic aneurysm repair: a secondary analysis from a prospective cohort study. Can J Anaesth. 2021 Dec;68(12):1756-1768. doi: 10.1007/s12630-021-02110-2. Epub 2021 Sep 27. PMID 34570352
- [Derived] Wang Y, Goralski KB, Roberts DJ, Landry K, Issa ME, Sleno L, Julien LC, Wood J, Hall RI. An observational study examining the effects of a surgically induced inflammatory response on the distribution of morphine and its metabolites into cerebrospinal fluid. Can J Anaesth. 2017 Oct;64(10):1009-1022. doi: 10.1007/s12630-017-0933-x. Epub 2017 Jul 14. PMID 28710563